CLINICAL TRIAL: NCT02601131
Title: Post-transfusion Platelet Count
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Thomas Kander, MD, PhD, Region Skane
Other Study IDs: Post-transf-PLC
Record Dates: First submitted 2015-10-28; First posted 2015-11-10 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Leukemia; Multiple Sclerosis
Keywords: platelet count; platelet transfusion; complement factors; endothelial markers; stem cell transplantation
MeSH Terms: conditions — Leukemia; Multiple Sclerosis | interventions — Platelet Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pending the analyses of complement factors and endothelial markers plasma is stored in -80 degrees Celcius. All samples are destroyed after analyses.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- AML, ALL and MDS: Patients receiving intensive chemotherapy with diagnoses of acute myeloid leukemia (AML), acute lymphocytic leukemia (ALL) or myelodysplastic syndromes (MDS).
  Interventions: Biological: Platelet transfusion
- Autologous stem cell transplantation: Patients undergoing autologous stem cell transplantation
  Interventions: Biological: Platelet transfusion
- Allogeneic stem cell transplantation: Patients undergoing allogeneic stem cell transplantation including both myeloablative conditioning (MAC) and the reduced-intensity conditioning (RIC)
  Interventions: Biological: Platelet transfusion
- Platelet transfusion prophylaxis: Patients receiving platelet transfusion prophylaxis before the intervention, such as insertion of a central venous catheter or lumbar puncture
  Interventions: Biological: Platelet transfusion
- Control: Patients with AML, ALL or MDS that have low PLC (10-20 billion/L) and is not relevant for platelet transfusion. Samples taken in the same manner as in the other groups. Control is needed to rule out other causes of variation of the PLC than the platelet transfusion and thereby strengthen the causality between a given transfusion and increased PLC.

INTERVENTIONS:
Biological: Platelet transfusion
  Groups: AML, ALL and MDS; Allogeneic stem cell transplantation; Autologous stem cell transplantation; Platelet transfusion prophylaxis

SUMMARY:
The purpose of this study is to identify how the platelet count, complement system and endothelial markers are affected over time, after platelet transfusion in 4 different hematological patient groups.

DETAILED DESCRIPTION:
Patients who are hospitalized at the Clinic for Hematology Diseases at the Skåne University Hospital (SUS) in Lund, Sweden with a central venous catheter or port-a-cath and should receive platelet transfusion due to thrombocytopenia are asked to participate in the study. Some patients who are being considered for platelet transfusions on several occasions will be able to attend more than one time in this study. After signed informed consent blood samples are drawn from the central line before, immediately after and then approximately. 1, 4, 8, 16 and 24 hours following the platelet transfusion. The platelet count (PLC) will then be taken daily following 4 days.

Sample size. Data from previous studies (Norol-98) shows that the PLC after platelet transfusion rises by 33 ± 25 x109/L (mean ± SD) 12 hours post-transfusion in patients with acute myeloid leukemia or pre-conditioning prior to bone marrow transplantation. The investigators want to show the same rise in the PLC after 12 hours with 80% power and 5% alpha risk of error for each group resulting in the sample size 13 per group and a total of 65 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Clinic of Hematology Diseases, Skåne University Hospital, Lund, Sweden belonging to either of the groups described in paragraph 8 above and are prescribed platelet transfusion.

Exclusion Criteria:

* Patients with aplastic anemia or treatment with antithymocyte globulin (ATG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Clinic of Hematology Diseases, Skåne University Hospital, Lund, Sweden
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in platelet count after platelet transfusion | 4 days after platelet transfusion

SECONDARY OUTCOMES:
Change in concentrations of complement factors in plasma after platelet transfusion | 4 days after platelet transfusion
Change in concentrations of endothelial markers in plasma after platelet transfusion | 4 days after platelet transfusion
Change in concentrations of complement factors in platelet rich plasma after platelet transfusion | 4 days after platelet transfusion
Analysis of platelets in platelet transfusions given to patients included in the study | 4 days after platelet transfusion
  Flow cytometry of platelets in platelet transfusions given to patients included in the study

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kander, MD, PhD, Principal Investigator — Region Skåne
Locations (1):
- Region Skåne, Lund, Sweden

REFERENCES:
- [Background] Norol F, Bierling P, Roudot-Thoraval F, Le Coeur FF, Rieux C, Lavaux A, Kuentz M, Duedari N. Platelet transfusion: a dose-response study. Blood. 1998 Aug 15;92(4):1448-53. PMID 9694735
- [Derived] Akesson A, Ljungkvist M, Martin M, Blom AM, Klintman J, Schott U, Zetterberg E, Kander T. Biomarkers of Complement and Platelet Activation are not correlated with the One or Twenty-Four Hours Corrected Count Increments in Prophylactically Platelet Transfused Hematological Patients: a Prospective Cohort Study. Platelets. 2022 Apr 3;33(3):350-359. doi: 10.1080/09537104.2021.1942817. Epub 2021 Jul 2. PMID 34210243